CLINICAL TRIAL: NCT03187522
Title: An EU Post-Approval Registry of the TREO® Stent-Graft for Patients With Infrarenal Abdominal Aortic Aneurysms
Brief Title: An European Union (EU) Post-Approval Registry of the TREO® Stent-Graft
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Post Market Study terminated early due to the launch and subsequent incorporation of the study into the Terumo Aortic Endovascular Registry (TiGER-001).
Sponsor: Bolton Medical (Industry)
Collaborators: Bolton Medical Espana SLU (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP-0020-16
Record Dates: First submitted 2017-06-11; First posted 2017-06-15 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2020-06

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: AAA; Abdominal Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-center, post-market clinical follow-up, non-randomized registry of patients treated with the TREO stent-graft
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TREO Stent-Graft (Experimental): Patients who receive a TREO Abdominal Stent-Graft System
  Interventions: Device: TREO Stent-Graft System

INTERVENTIONS:
Device: TREO Stent-Graft System — The TREO® Stent-Graft is designed for use in the management of patients with AAAs and is composed of self-expanding nitinol stents sutured to polyester vascular graft fabric.

SUMMARY:
This is an EU sponsored trial and independent of the US trial registered under Clinicaltrials.gov ID NCT02009644.

The purpose of this registry is to gather clinical data on the safety and performance of the TREO Stent-Graft in patients with infrarenal abdominal aortic aneurysms. The registry is part of TREO's EU post-market surveillance plan providing long-term systematic clinical follow-up.

DETAILED DESCRIPTION:
This is a prospective, multicenter, post-market clinical follow-up, non-randomized registry of the TREO Stent-Graft. Subjects diagnosed with infrarenal aortic aneurysms and treated with the TREO Stent-Graft or TREO aorto-uni-iliac (AUI) device can be included into the registry. Pre-procedure baseline data will be gathered as well as post-procedure assessments prior to hospital discharge and one to three months and 1, 2, 3, 4, and 5-year post-implantation.

The objective of the registry is to assess the clinical results and health economics of the TREO device in a real-world population of patients with infrarenal abdominal aortic aneurysms (AAA).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Signed informed consent
* Willingness to comply with study follow-up
* Indication for elective endovascular repair
* Planned implantation of single Treo device system or aorto uni-iliac (AUI) device to include any auxiliary device components

Exclusion Criteria:

* Intolerance to contrast media
* Emergency procedure
* Chimneys or fenestrated device procedures
* Connective tissue disease (e.g., Marfan's syndrome)
* High probability of non-adherence to follow-up requirements
* Current participation in a concurrent trial that may confound study results
* Female of childbearing potential in whom pregnancy cannot be excluded
* Previous endovascular or surgical AAA repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Aneurysm-related mortality | 30 days post-procedure
Stroke (excluding transient ischemic attack) | 30 days post-procedure
Myocardial infarction | 30 days post-procedure
  Raised cardiac enzymes within 30 days of the procedure
Renal failure | 30 days post-procedure
  Renal failure requiring renal replacement therapy (excluding renal insufficiency)
Respiratory failure | 30 days post-procedure
  excluding chronic obstructive pulmonary disease or pulmonary complications)
Paraplegia | 30 days post-procedure
  (excluding paraparesis)
Bowel ischemia | 30 days post-procedure
  A restriction in blood supply to tissues in the bowels
Treated aneurysm rupture | 30 days post-procedure

SECONDARY OUTCOMES:
Major Adverse Events (MAE) at the follow-up time points | 30 days post-procedure
  MAE includes any of the following : Aneurysm-related mortality, Stroke (excluding transient ischemic attack), Myocardial infarction, Renal failure requiring renal replacement therapy (excluding renal insufficiency), Respiratory failure (excluding chronic obstructive pulmonary disease or pulmonary complications), Paraplegia (excluding paraparesis), Bowel ischemia, Treated aneurysm rupture
Limb Ischemia | 30 days post-procedure
  Rate of clinically-evident ischemia, subcategorized by embolism or thrombosis, tabulated by the frequency of major amputation.
Secondary procedures | 5 years
  Freedom from aneurysm-related secondary procedures through five years follow-up. A questionnaire will be conducted. Investigators are required to conduct a lesion and device assessment at each follow-up visit. All secondary procedures reported will be treated descriptively in terms of results.
Vascular access complications | Vascular access will be evaluated on day of index procedure (implant)
  Injuries to vessels as a result of the endovascular procedure.
Patient-reported quality of life (QOL) | One year follow-up
  Health outcomes using the EuroQol Five Dimensions Questionnaire (EQ-5D) standardized EuroQol instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Torsello, MD, PhD, Principal Investigator — Center of Vascular and Endovascular Surgery, Munster University Hospital
Locations (16):
- Belgium (3):
  - Imelda Hospital, Bonheiden
  - Imeldaziekenhuis, Bonheiden
  - AZ Sint Blasius, Dendermonde
- Germany (3):
  - Bonifatius Hospital, Lingen
  - University Clinic and St. Franziskus Hospital Muenster, Münster
  - University Hospital Tübingen, Tübingen
- Compensorio Sanitario Bolzano, Bolzano, Italy
- Netherlands (2):
  - UMC Groningen, Groningen
  - UMCU, Utrecht
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona
  - Complexo Hospitalario Universitario de Ourense, Ourense
- Switzerland (2):
  - Centro Vascolare Ticino, Ospedale Regionale di Lugano, Lugano
  - Civico, Ospedale Regionale, Lugano
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge University Hospitals, Cambridge
  - Manchester Royal Infirmary, Central Manchester University Hospitals, Manchester
  - John Radcliffe Hospital, Oxford University Hospitals, Oxford

IPD SHARING:
Plan to Share IPD: No